CLINICAL TRIAL: NCT03962595
Title: Assessment Of Patient Satisfaction Of Outpatient Care In The Multi-Disciplinary Breast Clinic- Linguistic Validation Study
Brief Title: Patient Satisfaction Survey (PSS) In Breast Clinic
Acronym: PSS
Status: Completed | Type: Observational
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, Dr. Tabassum Wadasadawala, Associate Professor, Radiation Oncology, Breast Services, Tata Memorial Centre
Other Study IDs: 1835
Record Dates: First submitted 2019-05-01; First posted 2019-05-24 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Patient satisfaction is the primary means of assessing the effectiveness of primary health care delivery. It helps in improving the quality of care by identifying and help resolving the potential problem areas. It assesses the effectiveness of the care provided and document the quality to accrediting organisations.In our institute, we have developed a patient satisfaction survey (PSS) questionnaire and have conducted a pilot study (Institutional review board approved) with fifty English speaking breast cancer patients receiving active cancer directed treatment in outpatient clinic, to evaluate the level of patient satisfaction in them. Therefore, we are now conducting a linguistic validation study using Hindi and Marathi PSS questionnaire to assess the overall level of patient satisfaction in a larger cohort of patients with diverse linguistic and economic background attending both general and private Outpatient Clinic.

The aim of the study is to evaluate the overall level of patient satisfaction and their satisfaction at various encounters in the multi-disciplinary Breast Clinic which can be helpful to improve various aspects of patient care delivery.

Methods:

All patients who have already sort primary consultation in surgical, medical and radiation oncology outpatient clinics for their treatment plan and have had their last consultation within the last one month will be screened for the study. The Patient Satisfaction Survey (PSS) questionnaire (in preferred language) will be administered independently by a clinical research student who is not directly involved in patient care. The PSS will be anonymous. It will be administered to patients in the out-patient clinics waiting area. Patients will be asked to complete 3 surveys: one each for surgical, medical and radiation oncology professionals. It will take approximately 12 months to enroll the required number of patients.

Sample size: Previous studies conducted in India and the pilot study conducted at Tata Memorial Hospital (TMH) with the PSS questionnaire have shown that approximately 70% of the patients are satisfied with the health care services. Assuming that the proportion of patients satisfied with the health services, when assessed by Hindi and Marathi PSS questionnaire will be ± 5% of 70%, i.e. between 65% to 75%, a sample size of 340 will be needed to produces a two-sided 95% confidence interval, which is determined by using Confidence Intervals Formula- Clopper-Pearson method.

Potential Impact of the Study

1. Knowledge of patient satisfaction in breast cancer patients belonging to diverse linguistic and socio-economic background will help in improving the quality of life of patients using appropriate resources and measures relevant to Indian context.
2. Awareness of patient dissatisfaction will help improve doctor patient relationship.
3. Awareness of patient dissatisfaction will help to identify problem areas and improve the care delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Women with histological confirmation of breast cancer.
2. Planned to receive multi-disciplinary curative active cancer directed treatment.
3. Aware of their diagnosis and treatment plan.
4. Willingness to participate in study.
5. Patient able to read and comprehend Hindi and Marathi. -

Exclusion Criteria:

1. Eastern Cooperative Oncology Group 4
2. Unable to read and fill the questionnaire -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients attending both Private and General out-patient clinic for consultation will constitute the target population of the study.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Linguistic validation of patient satisfaction survey (PSS) questionnaires in Hindi and Marathi. | 1 Year
  Scoring: For each of the rated 25 items, a score of 1-5 will be assigned. This gives a maximum score of 125 and a minimum score of 25. A score of 75 or above indicates that patient is satisfied with the care provided.
  Construct validity for the instrument will be assessed using Pearson's correlation between the items and scales (It-Sc i.e. convergent validity) and between scales (Sc-Sc i.e. discriminant validity). The correlation coefficient should be >0.4 and <0.7 for these respectively.
  Internal consistency (scale reliability) of the multi item questionnaires will be tested by Cronbach alpha coefficient. The internal consistency should be 0.70 or higher when scales are used for group comparisons.

SECONDARY OUTCOMES:
Proportion of patients having mean overall satisfaction score <70 | 1 Year
  The distribution of patients having low satisfaction score < 70 across surgical, medical and radiation oncology will be studied and the comments provided by patients will help understand the reasons related to low satisfaction.
To compare the level of overall patient satisfaction between paid and service patients: percentage of patients having overall score below 75 of the maximum 125 | 1Year
  The comments provided by patients will help understand the reasons related to low satisfaction and the difference between the two classes of patients will be known from the percentage of patients having overall score below 70 of the maximum 125

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Tabassum Wadasadawala, MBBS,MD,DNB, Principal Investigator — Associate Professor, Breast Services
Locations (1):
- Tata Memorial Centre, Mumbai, Maharashtra, India

REFERENCES:
- See also: Sitzia J, Wood N. Patient satisfaction: A review of issues and concepts. Social Science and Medicine. 1997;45(12):1829-43. — https://www.ncbi.nlm.nih.gov/pubmed/9447632
- See also: Mendoza Aldana J, Piechulek H, al-Sabir A. Client satisfaction and quality of health care in rural Bangladesh. Bulletin of the World Health Organization. 2001; 79:512-7. — https://www.ncbi.nlm.nih.gov/pubmed/11436472
- See also: Lis CG, Rodeghier M, Gupta D. Distribution and determinants of patient satisfaction in oncology: A review of the literature. Patient Preference and Adherence. 2009;(3):287- — https://www.ncbi.nlm.nih.gov/pubmed/19936172
- See also: Landen CN, Younger NO, Collins Sharp B a., Underwood PB. Cancer patients' satisfaction with physicians: Princess Margaret hospital satisfaction with doctor questionnaire results. American Journal of Obstetrics and Gynecology. 2003 May;188(5):1177-9. — https://www.ncbi.nlm.nih.gov/pubmed/12748470
- See also: Bergenmar M, Nylén U, Lidbrink E, Bergh J, Brandberg Y. Improvements in patient satisfaction at an outpatient clinic for patients with breast cancer. Acta oncologica (Stockholm, Sweden). 2006 Jan;45(5):550-8. — https://www.researchgate.net/publication/6922305_Improvements_in_patient_satisfaction_at_an_outpatient_clinic_for_patients_with_breast_cancer
- See also: Brown RF, Hill C, Burant CJ, Siminoff L A. Satisfaction of early breast cancer patients with discussions during initial oncology consultations with a medical oncologist. Psycho-oncology. 2009 Jan;18(1):42-9. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4839191/